CLINICAL TRIAL: NCT01070836
Title: JCV Antibody Program in Patients With Relapsing Multiple Sclerosis Receiving or Considering Treatment With Tysabri: STRATIFY-2
Brief Title: JC Virus Antibody Study of Participants With Relapsing Forms of MS Receiving Treatment With Natalizumab
Acronym: STRATIFY-2
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 101JC402
Record Dates: First submitted 2010-02-17; First posted 2010-02-18 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: JCV; Sample Collection; PML; Antibody
MeSH Terms: interventions — Natalizumab

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — Plasma, Serum, Urine, Whole Blood, Peripheral blood mononuclear cell (PBMC)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- natalizumab: US participants with relapsing MS receiving commercial natalizumab
  Interventions: Drug: natalizumab

INTERVENTIONS:
Drug: natalizumab — Administered as specified in the treatment arm
  Other Names: Tysabri; BG00002

SUMMARY:
The primary objective of this study is to demonstrate that the incidence of progressive multifocal Leukoencephalopathy (PML) in natalizumab-treated participants who do not have detectable antibodies to John Cunningham virus (JCV) (antibody negative) is lower than in participants who have detectable antibodies to JCV (antibody positive).

The secondary objectives of this study are to: Estimate the incidence of PML in natalizumab-treated participants who are anti-JCV antibody negative and anti-JCV antibody positive, based on a meta-analysis of data obtained from this study and other data sources; Define the prevalence of anti-JCV antibody in relapsing multiple sclerosis (MS) participants receiving natalizumab within the TYSABRI Outreach: United Commitment to Health (TOUCH) Prescribing Program; Determine changes in anti-JCV antibody status over time.

DETAILED DESCRIPTION:
No treatment is provided in this observational, longitudinal cohort study. Study population will consist of United States (US) participants with relapsing MS receiving commercial natalizumab. There are no study-mandated visits. Serum samples will be collected during routine patient care or follow-up visits and will be sent to a central laboratory for analysis (presence of anti-JCV antibody), and remaining serum aliquots will be stored for future natalizumab and PML research. Additional samples will be collected at participating sites from participants who qualify and consent to participate in focused sampling group (participants who are anti-JCV antibody positive at any time point AND have received ≥12 infusions of natalizumab, whether or not they have a history of immunosuppressant use). These samples will be stored for future natalizumab and PML research.

ELIGIBILITY:
Key Inclusion Criteria:

* Relapsing MS patients receiving commercial natalizumab
* Patients receiving natalizumab and their prescribers must be enrolled in the TOUCH Prescribing Program.
* Patients with suspected or confirmed PML who are at or referred to a participating STRATIFY-2 site may enroll into STRATIFY-2 for purposes of PML sample collection.

Key Exclusion Criteria:

- Patients may participate in any other clinical trial or study sponsored by Biogen Idec ; however, if the anti-JCV antibody test is included in the other clinical study and that study is performing a longitudinal analysis of those samples, the patient should withdraw from STRATIFY-2.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: US participants with relapsing MS receiving commercial natalizumab.
Sampling Method: Probability Sample
Enrollment: 35895 (Actual)
Dates: Start 2010-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Demonstrate that the incidence of PML in natalizumab-treated participants who do not have detectable antibodies to JC virus (JCV) (antibody negative) is lower than in patents who have detectable antibodies to JCV (antibody positive) | Up to 4 years

SECONDARY OUTCOMES:
Estimate the incidence of PML in natalizumab-treated participants who are anti-JCV antibody negative and anti-JCV antibody positive, based on a meta-analysis of data obtained from this study and other data sources | Up to 4 years
Define the prevalence of anti-JCV antibody in relapsing MS participants receiving natalizumab within the TOUCH Prescribing Program | Up to 4 years
Determine changes in anti-JCV antibody status over time | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (394):
- United States (389):
  - Research Site, Birmingham, Alabama
  - Research Site, Cullman, Alabama
  - Research Site, Tucaloosa, Alabama
  - Research Site, Anchorage, Alaska
  - Research Site, Flagstaff, Arizona
  - Research Site, Gilbert, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Scottsdale, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Fayetteville, Arkansas
  - Research Site, Little Rock, Arkansas
  - Research Site, Sherwood, Arkansas
  - Research Site, Auburn, California
  - Research Site, Berkeley, California
  - Research Site, Carmel, California
  - Research Site, Carmichael, California
  - Research Site, Fountain Valley, California
  - Research Site, Fresno, California
  - Research Site, Fullerton, California
  - Research Site, La Jolla, California
  - Research Site, Loma Linda, California
  - Research Site, Los Alamitos, California
  - Research Site, Los Angeles, California
  - Research Site, Marina del Rey, California
  - Research Site, Modesto, California
  - Research Site, Newport Beach, California
  - Research Site, Northridge, California
  - Research Site, Palo Alto, California
  - Research Site, Pasadena, California
  - Research Site, Redding, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, San Francisco, California
  - Research Site, Santa Barbara, California
  - Research Site, St. Helena, California
  - Research Site, Stanford, California
  - Research Site, Stockton, California
  - Research Site, Thousand Oaks, California
  - Research Site, Tracy, California
  - Research Site, Arvada, Colorado
  - Research Site, Aurora, Colorado
  - Research Site, Basalt, Colorado
  - Research Site, Centennial, Colorado
  - Research Site, Colorado Springs, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Fort Collins, Colorado
  - Research Site, Greeley, Colorado
  - Research Site, Parker, Colorado
  - Research Site, Pueblo, Colorado
  - Research Site, Danbury, Connecticut
  - Research Site, Derby, Connecticut
  - Research Site, Fairfield, Connecticut
  - Research Site, Hartford, Connecticut
  - Research Site, New Haven, Connecticut
  - Research Site, New London, Connecticut
  - Research Site, Norwich, Connecticut
  - Research Site, Dover, Delaware
  - Research Site, Newark, Delaware
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Bradenton, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Fort Walton Beach, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Jacksonville Beach, Florida
  - Research Site, Lighthouse PT, Florida
  - Research Site, Maitland, Florida
  - Research Site, Melbourne, Florida
  - Research Site, Miami, Florida
  - Research Site, Naples, Florida
  - Research Site, Ocala, Florida
  - Research Site, Orange Park, Florida
  - Research Site, Orlando, Florida
  - Research Site, Ormond Beach, Florida
  - Research Site, Palm Bay, Florida
  - Research Site, Palm Beach Gardens, Florida
  - Research Site, Pompano Beach, Florida
  - Research Site, Ponte Vedra Beach, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Sarasota, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Sunrise, Florida
  - Research Site, Tallahassee, Florida
  - Research Site, Tampa, Florida
  - Research Site, Vero Beach, Florida
  - Research Site, Winter Haven, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Athens, Georgia
  - Research Site, Atlanta, Georgia
  - Research Site, Columbus, Georgia
  - Research Site, Johns Creek, Georgia
  - Research Site, Macon, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Snellville, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, Boise, Idaho
  - Research Site, Idaho Falls, Idaho
  - Research Site, Meridian, Idaho
  - Research Site, Nampa, Idaho
  - Research Site, Bloomington, Illinois
  - Research Site, Champaign, Illinois
  - Research Site, Chicago, Illinois
  - Research Site, Elk Grove Village, Illinois
  - Research Site, Elmhurst, Illinois
  - Research Site, Evanston, Illinois
  - Research Site, Flossmoor, Illinois
  - Research Site, Herrin, Illinois
  - Research Site, Lake Barrington, Illinois
  - Research Site, Lombard, Illinois
  - Research Site, Melrose Park, Illinois
  - Research Site, Niles, Illinois
  - Research Site, North Aurora, Illinois
  - Research Site, Palos Heights, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, St. Charles, Illinois
  - Research Site, Anderson, Indiana
  - Research Site, Bloomington, Indiana
  - Research Site, Elkhart, Indiana
  - Research Site, Evansville, Indiana
  - Research Site, Fort Wayne, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Lafayette, Indiana
  - Research Site, Merrillville, Indiana
  - Research Site, Mishawaka, Indiana
  - Research Site, Valparaiso, Indiana
  - Research Site, Ames, Iowa
  - Research Site, Des Moines, Iowa
  - Research Site, Iowa City, Iowa
  - Research Site, West Burlington, Iowa
  - Research Site, Hays, Kansas
  - Research Site, Kansas City, Kansas
  - Research Site, Lenexa, Kansas
  - Research Site, Overland Park, Kansas
  - Research Site, Topeka, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Paducah, Kentucky
  - Research Site, Alexandria, Louisiana
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Lacombe, Louisiana
  - Research Site, Lafayette, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Belfast, Maine
  - Research Site, Lewiston, Maine
  - Research Site, Scarborough, Maine
  - Research Site, Westbrook, Maine
  - Research Site, Annapolis, Maryland
  - Research Site, Baltimore, Maryland
  - Research Site, Bethesda, Maryland
  - Research Site, Frederick, Maryland
  - Research Site, Hagerstown, Maryland
  - Research Site, Attleboro, Massachusetts
  - Research Site, Boston, Massachusetts
  - Research Site, Brookline, Massachusetts
  - Research Site, Burlington, Massachusetts
  - Research Site, Milford, Massachusetts
  - Research Site, Peabody, Massachusetts
  - Research Site, Springfield, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Bingham Farms, Michigan
  - Research Site, Cinton Township, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, East Lansing, Michigan
  - Research Site, Farmington Hills, Michigan
  - Research Site, Grand Rapids, Michigan
  - Research Site, Kalamazoo, Michigan
  - Research Site, Midland, Michigan
  - Research Site, Muskegon, Michigan
  - Research Site, Rochester Hills, Michigan
  - Research Site, Roseville, Michigan
  - Research Site, Saginaw, Michigan
  - Research Site, Southfield, Michigan
  - Research Site, Traverse City, Michigan
  - Research Site, West Bloomfield, Michigan
  - Research Site, Woodhaven, Michigan
  - Research Site, Golden Valley, Minnesota
  - Research Site, Minneapolis, Minnesota
  - Research Site, Rochester, Minnesota
  - Research Site, Greenwood, Mississippi
  - Research Site, Hattiesburg, Mississippi
  - Research Site, Tupelo, Mississippi
  - Research Site, Kansas City, Missouri
  - Research Site, Nixa, Missouri
  - Research Site, Springfield, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Washington, Missouri
  - Research Site, Billings, Montana
  - Research Site, Great Falls, Montana
  - Research Site, Missoula, Montana
  - Research Site, Hastings, Nebraska
  - Research Site, Lincoln, Nebraska
  - Research Site, Norfolk, Nebraska
  - Research Site, North Platte, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Scottsbluff, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Reno, Nevada
  - Research Site, Lebanon, New Hampshire
  - Research Site, Bayonne, New Jersey
  - Research Site, Denville, New Jersey
  - Research Site, Edison, New Jersey
  - Research Site, Flemington, New Jersey
  - Research Site, Freehold, New Jersey
  - Research Site, Lawrenceville, New Jersey
  - Research Site, Livingston, New Jersey
  - Research Site, New Brunswick, New Jersey
  - Research Site, Newark, New Jersey
  - Research Site, Paterson, New Jersey
  - Research Site, Stratford, New Jersey
  - Research Site, Teaneck, New Jersey
  - Research Site, West Long Branch, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Albany, New York
  - Research Site, Amherst, New York
  - Research Site, Bay Shore, New York
  - Research Site, Brooklyn, New York
  - Research Site, Buffalo, New York
  - Research Site, Camillus, New York
  - Research Site, Cedarhurst, New York
  - Research Site, Corning, New York
  - Research Site, East Meadow, New York
  - Research Site, East Syracuse, New York
  - Research Site, Flushing, New York
  - Research Site, Fresh Meadows, New York
  - Research Site, Great Neck, New York
  - Research Site, Kingston, New York
  - Research Site, Lake Success, New York
  - Research Site, Latham, New York
  - Research Site, Mineola, New York
  - Research Site, Mount Kisco, New York
  - Research Site, New Hyde Park, New York
  - Research Site, New York, New York
  - Research Site, Newark, New York
  - Research Site, Patchogue, New York
  - Research Site, Plainview, New York
  - Research Site, Poughkeepsie, New York
  - Research Site, Rochester, New York
  - Research Site, Rye Brook, New York
  - Research Site, Schenectady, New York
  - Research Site, Staten Island, New York
  - Research Site, Stony Brook, New York
  - Research Site, Syracuse, New York
  - Research Site, West Seneca, New York
  - Research Site, White Plains, New York
  - Research Site, Williamsville, New York
  - Research Site, Woodmere, New York
  - Research Site, Advance, North Carolina
  - Research Site, Asheville, North Carolina
  - Research Site, Boone, North Carolina
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Concord, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Greenville, North Carolina
  - Research Site, Henderson, North Carolina
  - Research Site, Hendersonville, North Carolina
  - Research Site, High Point, North Carolina
  - Research Site, Mooresville, North Carolina
  - Research Site, Pinehurst, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Salisbury, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Bismarck, North Dakota
  - Research Site, Fargo, North Dakota
  - Research Site, Grand Forks, North Dakota
  - Research Site, Akron, Ohio
  - Research Site, Bellevue, Ohio
  - Research Site, Canton, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Franklin, Ohio
  - Research Site, Gahanna, Ohio
  - Research Site, Newark, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Uniontown, Ohio
  - Research Site, Youngstown, Ohio
  - Research Site, Zanesville, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Bend, Oregon
  - Research Site, Clackamas, Oregon
  - Research Site, Corvallis, Oregon
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Roseburg, Oregon
  - Research Site, Tulatin, Oregon
  - Research Site, Abington, Pennsylvania
  - Research Site, Allentown, Pennsylvania
  - Research Site, Altoona, Pennsylvania
  - Research Site, Bethlehem, Pennsylvania
  - Research Site, Brackenridge, Pennsylvania
  - Research Site, Collegeville, Pennsylvania
  - Research Site, Danville, Pennsylvania
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Erie, Pennsylvania
  - Research Site, Greensburg, Pennsylvania
  - Research Site, Harrisburg, Pennsylvania
  - Research Site, Hershey, Pennsylvania
  - Research Site, Johnstown, Pennsylvania
  - Research Site, Lititz, Pennsylvania
  - Research Site, Meadowbrook, Pennsylvania
  - Research Site, Monaca, Pennsylvania
  - Research Site, Monroeville, Pennsylvania
  - Research Site, Paoli, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Sellersville, Pennsylvania
  - Research Site, Tarentum, Pennsylvania
  - Research Site, Upland, Pennsylvania
  - Research Site, Washington, Pennsylvania
  - Research Site, West Reading, Pennsylvania
  - Research Site, York, Pennsylvania
  - Research Site, East Providence, Rhode Island
  - Research Site, Providence, Rhode Island
  - Research Site, Columbia, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Port Royal, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Bartlett, Tennessee
  - Research Site, Chattanooga, Tennessee
  - Research Site, Columbia, Tennessee
  - Research Site, Franklin, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Amarillo, Texas
  - Research Site, Arlington, Texas
  - Research Site, Austin, Texas
  - Research Site, Bedford, Texas
  - Research Site, Colleyville, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Kerrville, Texas
  - Research Site, Mansfield, Texas
  - Research Site, Round Rock, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Wichita Falls, Texas
  - Research Site, Ivins, Utah
  - Research Site, Provo, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, Washington Terrace, Utah
  - Research Site, Burlington, Vermont
  - Research Site, Alexandria, Virginia
  - Research Site, Carrollton, Virginia
  - Research Site, Centreville, Virginia
  - Research Site, Charlottesville, Virginia
  - Research Site, Christiansburg, Virginia
  - Research Site, Fairfax, Virginia
  - Research Site, Fredericksburg, Virginia
  - Research Site, McLean, Virginia
  - Research Site, Newport News, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Roanoke, Virginia
  - Research Site, Stafford, Virginia
  - Research Site, Vienna, Virginia
  - Research Site, Winchester, Virginia
  - Research Site, Auburn, Washington
  - Research Site, Bellingham, Washington
  - Research Site, Burien, Washington
  - Research Site, Federal Way, Washington
  - Research Site, Kirkland, Washington
  - Research Site, Mount Vernon, Washington
  - Research Site, Renton, Washington
  - Research Site, Richland, Washington
  - Research Site, Seattle, Washington
  - Research Site, Silverdale, Washington
  - Research Site, Spokane, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Wenatchee, Washington
  - Research Site, Huntington, West Virginia
  - Research Site, Point Pleasant, West Virginia
  - Research Site, Green Bay, Wisconsin
  - Research Site, La Crosse, Wisconsin
  - Research Site, Madison, Wisconsin
  - Research Site, Milwaukee, Wisconsin
  - Research Site, Neenah, Wisconsin
  - Research Site, Waukesha, Wisconsin
  - Research Site, Cheyenne, Wyoming
- Puerto Rico (5):
  - Research Site, Arecibo
  - Research Site, Bayamón
  - Research Site, Guaynabo
  - Research Site, Mayagüez
  - Research Site, Ponce